CLINICAL TRIAL: NCT01546012
Title: Assessment of Patient's Satisfaction Regarding the Handiness of Two Hyaluronic Acid Eye Drops Vials
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Too difficult to select patient according to the investigator
Sponsor: Laboratoires Thea (Industry)
Collaborators: Axial Biotech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: LT1550-PIV-CE-10/11; 2012-001233-14 (EudraCT Number)
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Assess the Patient Feeling About the Handiness of Two Different Vials Used to Deliver Both, Unpreserved Hyaluronic Eye Drops

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HYABAK® (Experimental): Hyaluronic Acid eye drops CE marked, packaged in multidose ABAK® container (preservative free)
  Interventions: Device: HYABAK®
- HYLO-COMOD®: (Active Comparator): Hyaluronic Acid eye drops CE marked, packaged in multidose COMOD® container (preservative free)
  Interventions: Device: HYLO-COMOD®

INTERVENTIONS:
Device: HYABAK® — Hyaluronic Acid eye drops CE marked, packaged in multidose ABAK® container (preservative free)
  Arms: HYABAK®
Device: HYLO-COMOD® — Hyaluronic Acid eye drops CE marked, packaged in multidose COMOD® container (preservative free)
  Arms: HYLO-COMOD®:

SUMMARY:
Assess the patient feeling about the handiness of two different vials used to deliver both, unpreserved hyaluronic eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 and older
* Patient with dry eye for at least 3 months
* Having given his written informed consent

Exclusion Criteria:

* Intolerance to studied products
* Patient's inability to understand the study procedures and give informed consent.
* Patient unwilling to follow the study procedures and visits defined by the protocol.
* Pregnant or lactating women.
* Patient under guardian ship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Overall preference of the patient | 6 weeks
  At Visit2: Week 6 +/- 1week: End of Study Visit. "Overall preference of the patient": number of answers Hyabak, Hylo-comod.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Erb, Principal Investigator — Augenklinik, Wittenbergplatz, Kleiststrasse 23-26, 10787 Berlin
Locations (1):
- Augenklinik, Berlin, Germany